CLINICAL TRIAL: NCT04063943
Title: Long-Term Follow-up of the Sidus® Stem-Free Shoulder Arthroplasty System
Brief Title: Long Term Sidus PMCF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has decided there is not a business need for this study and is not required to complete.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2018-27E
Record Dates: First submitted 2019-07-02; First posted 2019-08-21 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis; Post-traumatic; Arthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sidus Stem-Free Total Shoulder (Experimental): This arm will include all subjects who are implanted with the Sidus Stem-Free Total Shoulder Arthroplasty System
  Interventions: Device: Sidus Stem-Free Shoulder

INTERVENTIONS:
Device: Sidus Stem-Free Shoulder — Device: Sidus Stem-Free Total Shoulder Arthroplasty System

SUMMARY:
The objectives of this study are to assess the safety and performance of the Sidus Stem-Free Shoulder Arthroplasty System in unilateral primary total shoulder arthroplasty.

DETAILED DESCRIPTION:
The data collected from this study will serve the purpose of assessing safety and performance of the Sidus Shoulder.

Safety: Will be assessed by monitoring the frequency and incidence of adverse events (AE), serious adverse events (SAE), and unanticipated adverse device effects (UADE).

Performance: Will be determined by analyzing the implant survival, overall pain and functional performances (based on the ASES Patient Questionnaire and range of motion) and radiographic parameters of subjects who received the Sidus Shoulder. Implant survival will be based on removal or intended removal and determined using the observed component years (OCY) model as it is not anticipated that there will be adequate data at the 10 years follow-up to support Kaplan-Meier survivorship analysis. In the instance that there is sufficient data to perform Kaplan-Meier analysis, the analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have previously participated in the Sidus IDE clinical trial.
* Patient must not have undergone revision of the Sidus shoulder.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must be able and willing to sign the IRB/EC approved informed consent.

Exclusion Criteria:

* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient did not previously participate in the Sidus IDE clinical trial.
* Patient no longer has Sidus shoulder implanted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Safety: Monitoring frequency of AE, SAE and UADEs. | 10 Years
  Will be assessed by monitoring the frequency and incidence of adverse events (AE), serious adverse events (SAE), and unanticipated adverse device effects (UADE).
Performance: ASES Scores | 10 Years
  Will be determined by analyzing the ASES Questionnaire in subjects who received the Sidus Shoulder. ASES consists of 3 subcomponent scores including pain, instability and activities of daily living. The pain score can be 0 to 10 with 0 being no pain and 10 being the worst pain imaginable. The instability score can be 0 to 10 with 0 being no instability and 10 being the worst instability imaginable. The activities of daily living consists of 10 questions with ordinal responses of 0, 1, 2, and 3. 3 involves no limitation and 0 is unable to do. The 3 subcomponents combine to make the overall ASES score which can range from 0 to 100 with 0 being the worst possible score and 100 being the best.
Implant Survival | 10 Years
  Based on removal or intended removal of the device and determined using the OCY or Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN MBA, Study Director — Zimmer Biomet
Locations (7):
- United States (4):
  - Norton Orthopaedic & Sports Medicine, Louisville, Kentucky
  - MedStar Health, Baltimore, Maryland
  - Rothman Institute, Philadelphia, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania
- Canada (3):
  - University of Calgary Sports Medicine Clinic, Calgary, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - St. Joseph's Health Care London - Hand and Upper Limb Centre, London, Ontario